CLINICAL TRIAL: NCT03746041
Title: A Phase I Pilot Study of Abaloparatide + Bevacizumab in Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jason Mendler, Associate Professor of Hematology/Oncology, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00003054
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia
Keywords: Myelodysplastic syndromes; MDS; Chronic myelomonocytic leukemia; CMML; abaloparatide; bevacizumab; phase 1
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — abaloparatide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- abaloparatide and bevacizumab treatment (Experimental): In cycle 1, patients will be treated with single-agent, subcutaneous (SQ) abaloparatide at a dose of 80 mcg/day for 28 days. In cycles 2-4 (each cycle is 28 days), patients will be treated with SQ abaloparatide at a dose of 80 mcg/day and intravenous (IV) bevacizumab 5 mg/kg on days 1 and 15.
  Interventions: Drug: abaloparatide; Drug: bevacizumab

INTERVENTIONS:
Drug: abaloparatide — In cycle 1, patients will be treated with single-agent, subcutaneous (SQ) abaloparatide at a dose of 80 mcg/day for 28 days.
Drug: bevacizumab — In cycles 2-4 (each cycle is 28 days), patients will be treated with SQ abaloparatide at a dose of 80 mcg/day and intravenous (IV) bevacizumab 5 mg/kg on days 1 and 15.

SUMMARY:
The primary objective of this study is to determine the safety and tolerability of combined abaloparatide and bevacizumab in patients with Myelodysplastic Syndromes (MDS). A secondary objective is to determine the response to treatment (based on bone marrow and peripheral blood findings). A tertiary objective is to determine the impact of therapy on health-related quality of life (HRQOL) and patient-reported outcomes (PRO). A quaternary (scientific) objective is to determine the impact of treatment on both hematopoietic and stromal cell populations within the bone marrow of MDS patients.

DETAILED DESCRIPTION:
The main objective of this study is to determine the safety and tolerability of combined abaloparatide + bevacizumab in MDS patients. This will be a single center, single arm, phase 1 trial in MDS patients. In cycle 1, patients will be treated with single-agent, subcutaneous (SQ) abaloparatide at a dose of 80 mcg/day for 28 days. This will enable the investigator to monitor for any potential toxicities of single-agent abaloparatide in the MDS patient population. Following cycle 1, patients will have a bone marrow aspirate to determine the impact of abaloparatide treatment on bone marrow stromal cell and hematopoietic cell populations. In cycles 2-4 (each cycle is 28 days), patients will be treated with SQ abaloparatide at a dose of 80 mcg/day and intravenous (IV) bevacizumab 5 mg/kg on days 1 and 15. At the end of study, patients will have a bone marrow aspirate and biopsy to assess disease response and to determine the impact of combined abaloparatide + bevacizumab on bone marrow stromal cell and hematopoietic cell populations. After completion of trial therapy, another bone marrow aspirate and biopsy will be done 3 months later to assess the delayed impact of treatment. The investigator has chosen a phase 1 trial design because this combination has not been previously evaluated for toxicity. Since safe and effective doses of both abaloparatide and bevacizumab have already been identified and both drugs are Food and Drug Administration (FDA)-approved, the investigator does not feel there is a need to dose-escalate. The investigator will carefully monitor for therapy-limiting toxicities (TLTs) throughout the course of the study and impose an early stopping rule for toxicity. To monitor for TLTs, patients will have laboratory tests weekly and clinic visits every other week throughout the course of the trial. TLT is defined in the protocol with grading of adverse events defined by the NCI Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0. Response will be defined according to 2006 IWG working criteria for MDS. Patients who have achieved complete remission (CR), partial remission (PR), marrow CR, and/or hematologic improvement at any time during the 7 month trial period will be considered responders. Eligible subjects will have a diagnosis of MDS or non-proliferative chronic myelomonocytic leukemia (CMML) based on 2016 world health organization (WHO) criteria, and associated signs of bone marrow failure characterized by at least some degree of cytopenia involving at least one cell line such as anemia, thrombocytopenia or leukopenia. Patients will not be allowed to receive concurrent active chemotherapy or growth factors.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18
* Patients must have a documented diagnosis of MDS or non-proliferative chronic myelomonocytic leukemia (CMML) (WBC < 12,000/mcL) according to World Health Organization (WHO) criteria (27)
* Patients can be treatment-naïve or have received prior MDS-directed chemotherapy.

  * Treatment-naïve MDS patients (or those previously treated with growth factors alone) must have Revised International Prognostic Scoring System (IPSS-R) categories of Very Low-, Low- or Intermediate-risk disease (see Appendix A for Revised International Prognostic Scoring System for MDS).
  * MDS patients previously treated with disease-modifying chemotherapy (i.e. azacitidine, decitabine, lenalidomide, intensive chemotherapy, and/or an investigational agent) are eligible irrespective of IPSS-R score.
* Patients must be off all non-transfusion therapy for MDS for 28 days prior to initiation of study treatment, including all types of growth factors.
* Bone marrow biopsy (BMBx) within 30 days prior to first study treatment.
* Cytopenia involving at least one cell line such as anemia, thrombocytopenia or leukopenia at the time of study enrollment. Cytopenias should be present on at least 2 different blood draws within 8 weeks of study enrollment. Definitions of cytopenias for the purposes of this study are as follows:

  * Anemia: Patients must be symptomatic in the opinion of the treating physician with a hemoglobin ≤ 10.0 g/dL
  * Thrombocytopenia: Platelet count < 100,000/microliter
  * Neutropenia: Absolute neutrophil count < 1000/microliter
* ECOG Performance Status 0-2
* Adequate organ function as evidenced by:

  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × the upper limit of normal (ULN).
  * Total bilirubin ≤2 mg/dL
  * Serum creatinine <2 mg/dL, or creatinine clearance (calculated by the Cockcroft-Gault formula) ≤1.5 × ULN.
* Urine dipstick for proteinuria < 2+. Patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1 g of protein in 24 hours
* International normalised ratio (INR) ≤1.5 and prothrombin time (PT) ≤ 1.5 x ULN
* Women with an intact uterus (unless amenorrheic for the last 24 months) must have a negative serum pregnancy test within 30 days prior to enrollment into the study.
* Females of childbearing potential and sexually active males must use effective contraception during the trial and for 6 months after the last dose of bevacizumab.
* Written informed consent.

Exclusion Criteria:

* Bone marrow blasts equal to or greater than 20%
* Patients actively receiving either abaloparatide, teriparatide or bisphosphonate therapy for other indications
* Cumulative prior use of abaloparatide and/or any other parathyroid hormone analogs for > 20 months
* History of allogeneic stem cell transplant
* Pregnant or breast feeding female subjects
* Platelets < 50,000/mm3
* Major surgery (including open biopsy), significant traumatic injury within 28 days prior to enrollment or anticipation of the need for major surgery during study treatment
* Prior malignancy (excluding localized cervical carcinoma or cutaneous basal cell/squamous cell carcinoma) unless in remission for at least 2 years.
* Concurrent malignancy (excluding localized cervical carcinoma or cutaneous basal cell/squamous cell carcinoma)
* Need for aspirin at a dose of ≥ 325 mg/day; if aspirin can be safely stopped or dose dropped to < 325 mg/day ≥ 10 days before the first dose of bevacizumab, then patient will remain eligible
* Uncontrolled hypertension (blood pressures: systolic > 150 mmHg and/or diastolic > 100 mmHg)
* Clinically significant cardiovascular disease present ≤6 months before enrollment as judged by the treating physician. Examples include:

  1. Myocardial infarction
  2. Unstable angina
  3. Congestive heart failure NYHA Class ≥ II
  4. Serious cardiac arrhythmia
  5. Cerebrovascular accident and/or transient ischemic attack
  6. Severe peripheral vascular disease (ischemic rest pain, non-healing wound or ulcer, or tissue loss)
* Pulmonary embolus, deep venous thrombosis, or arterial thrombosis currently requiring anticoagulation
* < 10 days since prior anticoagulants
* Non-healing wound, active peptic ulcer or bone fracture
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months of enrollment
* Clinically significant hemorrhagic illness within the past 3 weeks
* History of osteosarcoma
* History of hyperparathyroidism
* Elevated (>ULN) serum calcium level
* Patients at increased risk for osteosarcoma, including those with Paget's disease of bone, unexplained elevations of alkaline phosphatase, and/or prior external beam or implant radiation therapy involving the skeleton.
* Psychiatric illness or social situation that would preclude study compliance
* Patients unable to give informed consent or to be followed up adequately
* Known hypersensitivity to a product from Chinese Hamster Ovary mammalian cell or to a recombinant humanized monoclonal antibody
* Other investigational treatments within 28 days of the start of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who experience a therapy-limiting Toxicity (TLT) | 7 months
  Safety of this therapy will be based on subjects who complete at least two cycles, experiencing both study drugs for at least one cycle. TLT is defined as any serious AEs considered at least possibly due to abaloparatide and/or bevacizumab, occurring at any time from the initial dose of study treatment, with severity graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.

SECONDARY OUTCOMES:
Proportion of patients who responded to therapy | 7 months
  In this study, patients who have achieved complete remission (CR), partial remission (PR), marrow CR, and/or hematologic improvement will be considered responders according to the International Working Group (IWG) Response Criteria and Modified IWG Response Criteria for Hematological Improvement. The overall rate of response will be estimated among all subjects who received at least one dose of any study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Mendler, M.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States